CLINICAL TRIAL: NCT02291705
Title: Ultrasound-guided Rectus Sheath Block In Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USG12
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain
Keywords: Ultrasound, rectus sheath block, children, inguinal hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Tramadol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rectus sheath block (Experimental): rectus sheath block
  Interventions: Procedure: rectus sheath block
- tramadol (Active Comparator): tramadol control group
  Interventions: Drug: Tramadol

INTERVENTIONS:
Procedure: rectus sheath block — ultrasound-guided rectus sheath block with 0.25% 0.2 ml/kg levobupivacaine
  Arms: rectus sheath block
Drug: Tramadol — tramadol 1 mg/kg iv
  Arms: tramadol

SUMMARY:
Inguinal hernia repair is one of the common day-case surgery in children. The aim of this study is to compare the effects of ultrasound guided rectus sheath block and intravenous tramadol on peroperative anesthetic requirement and postoperative analgesia.

DETAILED DESCRIPTION:
After approval the faculty ethical committee and informed consent from the parents (legal guardian) forty children aged 2-7 years scheduled for inguinal hernia repair were included in this prospective, randomized study. The patients were divided into two groups. After induction of general anesthesia, ultrasound guided rectus sheath block was applied to Group R with 0.2 mL/kg levobupivacain 0.25%. Tramadol 1 mg/kg intravenously was given to Group T before closure of the fascia. Intraoperative and postoperative hemodynamic parametres, postoperative pain by means of the FLACC were evaluated.

Primary end point was pain score using FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

* The children aged 2-7 years scheduled for inguinal hernia repair

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification III or greater, history of long term analgesic use, use of any analgesic within 24 hours before surgery, bleeding disorder, infection of application area, ultrasound imaging was inadequate and inability of the FLACC pain scoring system, substance sensitivity to local anesthetics.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain Scores | postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: dilek ozcengiz, MD, Study Director — CUKUROVA UNİVERSİTY
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Breschan C, Jost R, Stettner H, Feigl G, Semmelrock S, Graf G, Likar R. Ultrasound-guided rectus sheath block for pyloromyotomy in infants: a retrospective analysis of a case series. Paediatr Anaesth. 2013 Dec;23(12):1199-204. doi: 10.1111/pan.12267. Epub 2013 Sep 25. PMID 24112798
- [Background] Flack SH, Martin LD, Walker BJ, Bosenberg AT, Helmers LD, Goldin AB, Haberkern CM. Ultrasound-guided rectus sheath block or wound infiltration in children: a randomized blinded study of analgesia and bupivacaine absorption. Paediatr Anaesth. 2014 Sep;24(9):968-73. doi: 10.1111/pan.12438. Epub 2014 May 22. PMID 24853314
- [Background] Alsaeed AH, Thallaj A, Khalil N, Almutaq N, Aljazaeri A. Ultrasound-guided rectus sheath block in children with umbilical hernia: Case series. Saudi J Anaesth. 2013 Oct;7(4):432-5. doi: 10.4103/1658-354X.121079. PMID 24348296